CLINICAL TRIAL: NCT04364152
Title: Effects of Attentional Focus Strategy on Dual-task Walking Training in Parkinson's Disease With and Without Freezing of Gait
Brief Title: Effects of Attentional Focus Strategy on Dual-task Walking Training in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202001029RIND
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease; Dual-task Walking
Keywords: Parkinson; dual-task training; attention; electroencephalogram (EEG)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PD patients with freezing of gait, internal strategies (Experimental): Participants in this group will include PD patients with freezing of gait. During dual-task walking training, internal attentional strategies will be given, aiming to improve their gait performance.
  Interventions: Behavioral: Dual-task walking training
- PD patients with freezing of gait, external strategies (Experimental): Participants in this group will include PD patients with freezing of gait. During dual-task walking training, external attentional strategies will be given, aiming to improve their gait performance.
  Interventions: Behavioral: Dual-task walking training
- PD patients without freezing of gait, internal strategies (Experimental): Participants in this group will include PD patients without freezing of gait. During dual-task walking training, internal attentional strategies will be given, aiming to improve their gait performance.
  Interventions: Behavioral: Dual-task walking training
- PD patients without freezing of gait, external strategies (Experimental): Participants in this group will include PD patients without freezing of gait. During dual-task walking training, external attentional strategies will be given, aiming to improve their gait performance.
  Interventions: Behavioral: Dual-task walking training
- Healthy elders, internal strategies (Experimental): Participants in this group will include healthy elders. During dual-task walking training, internal attentional strategies will be given, aiming to improve their gait performance.
  Interventions: Behavioral: Dual-task walking training
- Healthy elders, external strategies (Experimental): Participants in this group will include healthy elders. During dual-task walking training, internal attentional strategies will be given, aiming to improve their gait performance.
  Interventions: Behavioral: Dual-task walking training

INTERVENTIONS:
Behavioral: Dual-task walking training — Participants will be instructed to perform both motor and cognitive dual-task walking during exercise training. For example, for motor dual-task walking, the participants may be instructed to throw and catch a ball while walking. As for cognitive dual-task walking, the participants may be instructed to name animals or perform calculation while walking.

SUMMARY:
Walking deficits and altered brain capacity have been proved to be two of the main contributing factors in dual-task walking deficits in patients with Parkinson's disease (PD). In the past, patients with PD were usually suggested not to walk in dual-task conditions in order to concentrate on their walking performance better. However, since dual-task walking is really common in daily-life, this limitation usually lead to a decrease in quality of life for PD patients. In previous studies, effects of using attentional strategies in dual-task walking training remain unclear, while suitable attentional strategies and corresponded neuroplasticity for patients with and without freezing of gait have not been well discussed, either. Accordingly, this study is aimed to identify (1) whether internal or external attentional strategies is more ideal for PD patients with and without freezing of gait in dual-task walking training, and (2) changes in brain activity after receiving dual-task walking training with different attentional strategies in patients with or without freezing of gait. Our hypothesis are (1) patients with or without freezing of gait will react differently in dual-gait training with different attentional strategies, and (2) changes in brain activities will be different according to different attentional strategies given in the training.

DETAILED DESCRIPTION:
The hypothesis will be tested by gait performance, suprapostural tasks performance, relative power spectrum of EEG, and scales including MDS-UPDRS, ABC, BBS, and TUG.

ELIGIBILITY:
Inclusion Criteria:

for PD patients:

* (1) a diagnosis of idiopathic PD by a neurologist expert in movement disorders (2) onset age > 40 years old, (3) presence of gait disorders or freezing of gait (points on 3.10 in MDS-UPDRS>=1 or points on item 3 in NFOG-Q >0) (4) able to walk independently without an assistance device at least for 20 meters (5) without obvious action or postural tremor, according to the score of 3.15 and 3.16 (action and postural tremor of hands) in MDS-UPDRS

for healthy elders:

* (1) without musculoskeletal of neurological diseases which may affect balance or walking performance (2) no medication that might influence their balance or cognition (3) MMSE> 26 points.

Exclusion Criteria:

for PD patients:

* (1) with other neurological or musculoskeletal disease that might affect balance or walking (2) have a Mini-Mental State Examination (MMSE) < 27 points (3) have a history of brain surgery (4) have to modulate their medication for duration of the experiment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Gait velocity from GAITRite | 60 minutes
  gait performance
Cadence from GAITRite | 60 minutes
  gait performance
Mean step length from GAITRite | 60 minutes
  gait performance
Step-to-step variability from GAITRite | 60 minutes
  gait performance
Amplitude from a triaxial accelerometer, X axes | 25 minutes
  motor suprapostural task performance
Amplitude from a triaxial accelerometer, Y axes | 25 minutes
  motor suprapostural task performance
Amplitude from a triaxial accelerometer, Z axes | 25 minutes
  motor suprapostural task performance
Correct rate on working memory task | 25 minutes
  cognitive suprapostural task performance

SECONDARY OUTCOMES:
EEG relative power in the delta band | 60 minutes
  brain activity under single, motor dual-task, and cognitive dual-task walking conditions
EEG relative power in the theta band | 60 minutes
  brain activity under single, motor dual-task, and cognitive dual-task walking conditions
EEG relative power in the alpha band | 60 minutes
  brain activity under single, motor dual-task, and cognitive dual-task walking conditions
EEG relative power in the beta band | 60 minutes
  brain activity under single, motor dual-task, and cognitive dual-task walking conditions
EEG relative power in the low gamma band | 60 minutes
  brain activity under single, motor dual-task, and cognitive dual-task walking conditions

CONTACTS AND LOCATIONS:
Locations (1):
- School and Graduate Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No